CLINICAL TRIAL: NCT03959904
Title: The Impact of Abdominal Wall Closure Technique on Incidence of Incisional Hernia in Kidney Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B00469
Record Dates: First submitted 2019-04-08; First posted 2019-05-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Surgery--Complications
MeSH Terms: interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Intervention Model Description: 2 groups randomised to different suturing techniques following surgery
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Stitch (Active Comparator): Small stitch for wound closure
  Interventions: Procedure: Small stitch; Other: Blood sample; Other: Tissue Sample; Other: Pain Score; Other: Quality of Life Score
- Large Stitch (Active Comparator): Large Stitch for wound closure
  Interventions: Procedure: Small stitch; Other: Blood sample; Other: Tissue Sample; Other: Pain Score; Other: Quality of Life Score

INTERVENTIONS:
Procedure: Small stitch — Wound closure will be using small stiches or larger spaced stitches
  Other Names: Large Stitch
Other: Blood sample — A blood sample to look for biological markers of Hernia formation will be taken
Other: Tissue Sample — A tissue sample will be taken to measure markers of wound healing.
Other: Pain Score — A pain score will be recorded following the surgical procedure.
Other: Quality of Life Score — A Quality of Life Score will be recorded at 1 month 6 months and 12 months post surgery

SUMMARY:
STUDY SUMMARY Incisional hernias, or swellings of the abdominal scar after surgery, remain problematic especially after transplant surgery. This is because they can cause complications, including trapping of bowel or the transplant. This can cause life threatening emergencies but is at the very least unsightly and uncomfortable for the patient. Transplant patients are especially likely to develop hernias because of the diseases causing the renal failure and the drugs that they take to dampen the immune system. There is evidence from other surgery that the stitching methods that are used to close the wounds might decrease the risk of surgical hernias. This is achieved by placing smaller and more numerous sutures (stitches) in the wound to increase the strength of the repair. However, this has never been tested formally in transplant where it may provide significant benefit. We intend to do some initial investigation of whether using the smaller stitches may provide benefit over more traditional methods that are currently being used. We will look at early complications after surgery but also the rate of hernia formation later. We hope to improve outcomes and reduce complications for our transplant patients by doing this. In addition we will collect blood and tissue samples from both live kidney donors and the recipients to microscopically analyse their collagen to identify potential factors which may indicate risk of hernia formation.

DETAILED DESCRIPTION:
Study Design This study has two phases. In phase 1 we will perform a retrospective review of hernia incidence in our centre over the last decade. We will seek to identify risk factors in our transplant cohort. In phase 2 we will perform a prospective randomised blinded feasibility trial in which the conventional large bites technique will be compared with the small bites technique.

STUDY SETTING The study will be carried out on one site at Manchester Royal Infirmary, part of Manchester University National Health Service (NHS) Foundation Trust. This is a regional Renal and Pancreas Transplant centre performing approximately 60 pancreas transplants per annum and 350 kidney transplants. All members of the team have academic track records and participate in several on-going research projects. Current research projects are investigating cardiovascular disease, kidney perfusion, Magnetic Resonance (MR) imaging to name a few.

RESEARCH QUESTIONS, AIMS, AND OBJECTIVES

Phase 1 To retrospectively evaluate the incidence of incisional hernias in our transplant population and associated risk factors.

Phase 2

1. To perform prospective randomized double blinded feasibility trial to investigate the use of "small bites" (SB) vs "large bites (LB)" for closure of abdominal incisions following kidney transplantation.
2. To collect detailed medical histories from all patients included in the study to look for potential medical risk factors which may predispose to hernia formation.
3. To collect tissue and blood samples to investigate potential biological and histological markers of hernia formation, from both patients with end stage renal failure receiving a living-donor kidney transplant, and samples from the donor nephrectomy patients for histological comparison.
4. To assess quality of life and pain scores in the early and delayed post-operative phase (week 1, 6 months and 1 year)

Outcomes Phase 1 Incidence of Incisional Hernia within 1 and 3 years post-transplant clinically or radiologically detected.

Phase 2 Primary outcome Incidence of Incisional Hernia within one year post transplant, either clinically or radiologically detected. Any incisional hernia identified will be classified as per European Hernia Society Guidelines.

Secondary outcomes Incidence of post-operative complications at 6 months post op (burst abdomen, chest infection, surgical site infection returns to theatre,etc), pain score, costs, length of hospital stay, quality of life at week 1, 6 and 12 months post-transplant, collagen and serum biomarkers which may predispose to hernia formation

Sampling and recruitment Sample identification Phase 1 Data will be collected from the medical records of our Transplant population and entered into an excel spreadsheet no personal identifiers will be recorded.

Phase 2 The Chief Investigator (CI) and Principle Investigator (PI) will identify patients on the transplant waiting list and send copies of the information sheet.

Following ethical approval, patients undergoing first or second renal transplantation will be asked for informed consent to participate in the study to receive either small or large bites.

The CI and PI are part of the direct care team. The CI will have custody of the clinical information.

Clinical details will be recorded on hospital pass worded computers. Blood samples will be anonymised at the time of collection. Patients will be given a study code and blood samples will be labelled with this code to ensure anonymity.

The custodian of the data and samples will be the CI.Mr David van Dellen.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal failure patients
* Aged 18-70yrs
* First transplants or second transplants
* Ability to adequately understand English and consent for study
* BMI<35 kg/m2)
* Living donor nephrectomy patients Exclusion Criteria
* Outside age range,
* Previous transplants which have left a scar in the ilia fossa

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hernia | 1 year
  Incidence of Incisional Hernia within one year post transplant, either clinically or radiologically detected. Any incisional hernia identified will be classified as per European Hernia Society Guidelines.

SECONDARY OUTCOMES:
Number of Complications | 1 year
  Incidence of post-operative complications at 6 months post op (burst abdomen, chest infection, surgical site infection, returns to theatre).
Pain Scores | 1 week 6 months and 12 months
  The level of pain as assessed by a pain score.
Length of Stay in Hospital following surgery | Number of days in hospital in 12 months post operation
  The number of days in hospital
Quality of Life Post surgery | 1 week 6 months 12 months post surgery
  A quality of life questionnaire will be administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No